CLINICAL TRIAL: NCT05103319
Title: Simultaneous Application of Ketamine and Lidocaine During an Ambulatory Infusion Therapy as a Treatment Option in Refractory Chronic Pain Conditions - A Retrospective Analysis
Brief Title: Simultaneous Application of Ketamine and Lidocaine During an Ambulatory Infusion Therapy as a Treatment Option in Refractory Chronic Pain Conditions
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01285; am21Schneider
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain
Keywords: lidocaine; ketamine
MeSH Terms: conditions — Chronic Pain | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection for statistical analysis to identify patterns of treatment response/ non-response — All data are restricted from the patient physical and electronic record of the Pain Management-Unit of the University Hospital Basel. No external data sources will be used. Records will be screened from 2012- May 2021. Variables collected are e.g. demography, medical diagnosis, psychological diagnosis, infusion therapy, medication, pain.

SUMMARY:
This study is to retrospective investigate the effects of the simultaneous intravenous (i.v.) administration of lidocaine and ketamine on a four to six weeks interval in treatment refractory different chronic pain conditions.

DETAILED DESCRIPTION:
The use of intravenous infusion therapy with lidocaine or ketamine has been of interest in several chronic pain conditions. Studies showed a benefit in immediate pain reduction and even longer lasting pain relief for treatment approaches with lidocaine and ketamine.

While there is a broad database on the use of lidocaine and ketamine in chronic pain management as separate agents, very few pre-clinical animal studies have investigated the combined use of said analgesics and none of them reports their combined use in chronic pain patients.

This study is to retrospective investigate the effects of the simultaneous i.v. administration of lidocaine and ketamine on a four to six weeks interval in treatment refractory different chronic pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* ICD11 Medical diagnosis of chronic pain and its subcategories
* Treatment with intravenous lidocaine and ketamine infusions during the years of 2012 to May 2021 at our pain unit at the USB
* Patient is at least 18 years of age at the beginning of the first infusion treatment

Exclusion Criteria:

* Patient is underage at the beginning of the first infusion treatment
* Documented written refusal of consent for research (general consent or specific study consent)
* Patients undergoing treatment with only lidocaine or ketamine respective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study only includes patients treated with lidocaine-ketamine infusions at the pain unit in the University Hospital of Basel (2012 -until May 2021) All data are extracted from the paper or electronic patient chart of the Pain Management-Unit of the University Hospital Basel. All data are collected retrospectively.
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction over time (long lasting) | up to 1 year
  The primary outcome (pain reduction over time) is explorative and not comparative, therefore no hypothesis is formulated and only descriptive/explorative statistics will be applied. Pain reduction will be analysed descriptively. Categories: any pain reduction/ pain reduction >=50%/ pain free/ increase in pain (recorded as "no time stated/ < 2 weeks/ ≥2 weeks/full time in-between infusions"

SECONDARY OUTCOMES:
Change in Pain (acute reduction) | up to 1 day
  Numeric rating scale (NRS) at start of infusion (recorded as number from 0 = no pain to 10 = maximal pain)/ NRS at end of infusion (recorded as number from 0 to 10)

OTHER OUTCOMES:
Change in activity | up to 1 year
  Categories: increased activity/ quantifiable increased activity/ activity without restrictions/ decreased activity (recorded as "no time stated/ < 2 weeks/ ≥2 weeks/full time in-between infusions" for each category)
Change in sleep | up to 1 year
  Categories: increased quality of sleep/ decreased quality of sleep (recorded as "no time stated/ < 2 weeks/ ≥2 weeks/full time in-between infusions" for each category)
Change in mood | up to 1 year
  Categories: mood brightened/ mood worsened (recorded as "no time stated/ < 2 weeks/ ≥2 weeks/full time in-between infusions" for each category)
Number of side effects | up to 1 year
  Categories: waking reactions such as hallucinations, vivid dreams, nightmares, confusion, fidgetiness, agitation/ raise in liver enzymes/ sight disorders, diplopia/ anxiety/ nystagmus, tonic and clonic movement, increased muscle tone, increased intracranial pressure/ dizziness/ tachycardia/ bradycardia/ hypertension/ hypotension/ respiratory depression/ nausea, vomiting/ erythema/ acute kidney impairment, hemorrhagic cystitis, hydronephrosis/ signs and symptom of cns toxicity (convulsions, paraesthesia circumoralis, numbness of tongue, hyperacusis, tremor, tinnitus, dysarthria, cns depression)
Change in medication | up to 1 year
  Categories: Substance name (recorded as free text)/ amount of substance at start (recorded in mg)/ date at start/ amount of substance after change (recorded in mg)/ date of change
Infusion therapy | up to 1 year
  Categories: Amount of infusions totally received (recorded as number)/ time frame of infusion therapy (date at beginning/ date at end)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Schneider, Dr. med., Principal Investigator — Department of Anesthesiology University of Basel (USB)
Locations (1):
- Department of Anesthesiology, University of Basel (USB), Basel, Switzerland

REFERENCES:
- [Derived] Striebel J, Ruppen W, Schneider T. Simultaneous application of lidocaine and ketamine during ambulatory infusion therapy: a retrospective analysis. Pain Manag. 2023 Sep;13(9):539-553. doi: 10.2217/pmt-2023-0037. Epub 2023 Oct 18. PMID 37850330